CLINICAL TRIAL: NCT04720989
Title: The Effect of Cleansing Product Used in the First Bathing on Transepidermal Water Loss and Skin Ph in Late Preterm and Term Infants: A Multicenter, Evaluative Blind Randomized Controlled Study
Brief Title: Cleanser Versus Only Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Research Assistant, Doctoral Candidate, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK-929
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Premature Birth
Keywords: Skin Barrier Function; First Bathing; Baby Cleanser; Transepidermal Water Loss; Skin pH
MeSH Terms: conditions — Premature Birth | interventions — Baths; Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing With Baby Cleanser (Experimental): Skin cleansing products will be used in the first baths of the participants in this group.
  Interventions: Procedure: Bathing With Baby Cleanser and water
- Bathing With only Water (Experimental): Only water will be used in the first baths of the participants in this group.
  Interventions: Procedure: Bathing With only Water

INTERVENTIONS:
Procedure: Bathing With Baby Cleanser and water — Late preterm and term newborns, whose informed consents are obtained by their parents to participate in the project, will be given their first baths according to the intervention group they are assigned to. Before the first bath / after birth, preterm newborns in all groups will be wiped only once with a clean towel without removing the vernix caseosa. Newborns who were bathed before the application of the study will be excluded from the study. As the most appropriate time for bath time, 30 minutes after the end of the feeding and treatment of the newborns, the bath application will be made at any time between 9 pm and 3 pm.
  Arms: Bathing With Baby Cleanser
Procedure: Bathing With only Water — Preterm infants will have their first baths only with water.
  Arms: Bathing With only Water

SUMMARY:
The aim of this study is to determine the effect of the newborn's first bath with a cleaning product and only water on the barrier function of the skin.

DETAILED DESCRIPTION:
Studies in the literature on the effects of newborn bath types on the effects of body temperature on newborn crying times, on the effects of newborn behavior and stress, the views and practices of mothers with newborn babies on baby bathing, and the effects of bath types on the umbilical cord in term babies, and the effects of bath products on newborns. It seems that there are studies done. However, although studies on the effect of the cleaning product used in the first bath of late preterm and term newborns on the skin barrier are limited in number for term newborns, there are almost no studies for late preterm newborns. The hypotheses of this study are as follows; 1. In late preterm and term newborns, the first bath with cleaning product protects the newborns' Transepidermal Fluid Loss better than the first bath with only water. 2. In late preterm and term newborns, the first bath with cleansing product keeps the skin pH levels of newborns at a more optimal level compared to the first bath with only water.

ELIGIBILITY:
Inclusion Criteria:

* Born between 34 weeks + 0 days and 42 weeks + 6 days (late preterm and term),
* With a body weight of 1800g or more,
* Spontaneous breathing,
* Preterms with stable physiological parameters will be included in the study.

Exclusion Criteria:

* Receiving mechanical ventilation support,
* Mother's baby with HIV, Hepatitis B,
* Preterms who had a bath before the intervention,
* Surgical operation and incision in any area,
* Preterms with a central catheter,
* Preterms with systemic infections,
* Preterms using sedatives and / or muscle relaxants,
* Preterms with congenital or chromosomal anomalies

Ages: 34 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Transepidermal Water Loss | Change from Baseline (10 minutes before first bathing) Transepidermal Water Loss at 10 minutes and 30 minutes after bathing.
  Among the outcome criteria, the skin barrier function will be evaluated first. Skin barrier function will be evaluated by measuring Transepidermal Water Loss (TESK). To measure transepidermal water loss, it will be measured by closed chamber evaporation using VapoMeter SWL-2 ™ (Delfin Technologies Ltd).

SECONDARY OUTCOMES:
Skin pH Level | Change from Baseline (10 minutes before first bathing) skin pH at 10 minutes and 30 minutes after bathing.
  In the secondary outcome measure of the research, results related to the skin pH level will be shown. Skincheck HI 98109 ™ will be used to measure these results.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Principal Investigator — http://hemsirelik.akdeniz.edu.tr/iletisim/
Locations (1):
- Akdeniz Universty, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If he/she wishes, he/she can be contacted after the broadcast stage.(eril)